CLINICAL TRIAL: NCT02449876
Title: The Feasibility of Using Neuroscience Education in Adults Over 65 Years Old With Chronic Low Back and/or Lower Extremity Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Adam Rufa, Clinical Assistant Professor, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNE 123
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Back Pain; Lower Extremity Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neuroscience Education (Experimental): Subjects will have 2 sessions of education 2 weeks apart. After the first session subjects will be given a 50 page book "Why Do I Hurt" by Adriaan Louw. Session 1 will last approximately 60 minutes and session approximately 30 minutes.
  Interventions: Other: Neuroscience Education

INTERVENTIONS:
Other: Neuroscience Education — The following topics will be discussed in the education
  * Basic structure of the nervous system
  * Basic physiology of the nervous system
  * The function and importance of pain
  * Strategies to lessen the impact of pain
  The instruction will be delivered in an interactive manner so that questions are addressed immediately. At the conclusion of the session each subject will receive the book: Why Do I Hurt by Adriaan Louw to reinforce the information discussed in the session. Subjects will be asked to read the 50 page book prior to the second session.
  Session 2:
  The session will begin with a review of the topics discussed in Session 1 and contained in the book. Subject will be encouraged to ask questions and get clarification on any of the topics that are unclear.
  Other Names: Therapeutic Neuroscience Education

SUMMARY:
This is a pilot study to determine if neuroscience education is acceptable to adults over 65 and if it can have an impact on pain, pain beliefs and gait speed

DETAILED DESCRIPTION:
Background: Health care professionals commonly provide education to patients who are in pain. Traditionally, this education has focused on pathoantaomical aspects of the patient's condition.(1,2) Despite the popularity of this type of education the evidence has indicated that it either has little effect (2-4) or in some cases can have a negative effect on pain and disability.(3,5-7) In contrast, therapeutic neuroscience education (TNE) directly addresses cognitions about pain by teaching patients basic pain physiology and addressing abnormal pain beliefs (e.g., pain=harm). TNE has been shown to produce positive changes in pain beliefs, including a reduction in pain catastrophizing, and improvements in both pain levels and pain-related disability. (2,3,8) To date, research on the impact of TNE has focused on working-aged adults. Pain however, is highly prevalent among the older adult population, leading to activity limitation and pain-related disability.(4-7) The purpose of this project is to determine whether older adults are receptive toTNE, if TNE can have an impact on the gait speed of older adults and if TNE can have an impact on pain beliefs.

Methods: This will be a single group, uncontoled pilot study of 15-20 adults aged 65 years and older who report low back or lower extremity pain. Subjects will be recurited from physician offices and the community via flyers and word of mouth. Subjects will be screened for eligibility and informed consent will be obtained. Inclusion criterion will include age over 65, self-reported back and/or lower extermity pain present on most days for at least three months, be independent with ambulation (with or without and assistive device) and English speaking. Exclusion criteria include cancer-related pain, recent (within 6 months) surgery on the back or lower extremities affecting mobility, current ongoing treatment by another healthcare professional for low back or lower extremity pain (including physical therapy, chiropractic or massage) or other diagnoses that impact mobility or rusult in cognitive limitations.

Upon enrollment in the study each subject will complete intake questionnaires (basic demographic information, the Tampa Scale of Kinesiophobia (TSK), Pain Disability Index (PDI), and Resilience Scale( RS), and one physical performance measure (Gait Speed, preferred and maximal).

The educational material will be delivered in two, one on one, meetings for a total time of approximately ninety minutes. The first meeting will last about one hour and all of the educational content will be delivered in this session. A supplemental handout (reference), which will highlight the concepts covered in the presentation, will be given to each subject. The second educational session will serve as a review of the material covered in the first meeting and described in the supplemental materials. During this session subjects will be encourage to ask questions and get clarification about any of the covered topics which are unclear. At the conclusion of the second session the surveys initially administered will be repeated (TKS, PDI, RS), the gait speed test will be repeated and a brief survey about the education will be administered.

1. Butler D, Moseley L, eds. Explain pain. Australia: NOI Group Publishing; 2003.
2. Brox JI, Storheim K, Grotle M, Tveito TH, Indahl A, Eriksen HR. Systematic review of back schools, brief education, and fear-avoidance training for chronic low back pain. Spine J. 2008;8(6):948-958.
3. Maier-Riehle B, Harter M. The effects of back schools--a meta-analysis. Int J Rehabil Res. 2001;24(3):199-206.
4. Koes BW, van Tulder MW, van der Windt WM, Bouter LM. The efficacy of back schools: A review of randomized clinical trials. J Clin Epidemiol. 1994;47(8):851-862.
5. Nachemson AL. Newest knowledge of low back pain. A critical look. Clin Orthop Relat Res. 1992;(279)(279):8-20.
6. Poiraudeau S, Rannou F, Baron G, et al. Fear-avoidance beliefs about back pain in patients with subacute low back pain. Pain. 2006;124(3):305-311.
7. Hirsch MS, Liebert RM. The physical and psychological experience of pain: The effects of labeling and cold pressor temperature on three pain measures in college women. Pain. 1998;77(1):41-48.
8. Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011;92(12):2041-2056.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years old, have low back and/or lower extremity pain present on most days for at least three months, be independent with ambulation (with or without assistive device) and English speaking.

Exclusion Criteria:

* cancer related pain, recent surgery (within 6 months) on the back or lower extremities affecting mobility, current ongoing treatment by another healthcare professional for low back or lower extremity pain (including physical therapy, chiropractic or massage) or the presence of other diagnoses that impact mobility or result in cognitive limitations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia | 2 weeks
Pain Disability Index | 2 weeks
Neuroscience education acceptance and understanding survey | 2 weeks
  Adapted from Louw 2013, Am J Phys. Med. Rehabil
Preferred and fast gait speed | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Human Performance, Syracuse, New York, United States